CLINICAL TRIAL: NCT06966830
Title: A Multicenter, Prospective, Real-World Observational Study of Lacosamide Intravenous Injection for Emergency Termination of Status Epilepticus
Brief Title: Lacosamide Intravenous Injection for Emergency Termination of Status Epilepticus
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: First Affiliated Hospital of Jinan University (Other); Guangzhou First People's Hospital (Other); Southern Medical University, China (Other); Guangdong 999 Brain Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-LCYJ-ZF-44
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Epilepsy; Status Epilepticus
Keywords: Lacosamide; Intravenous Injection; Emergency Termination; Efficacy
MeSH Terms: conditions — Epilepsy; Status Epilepticus | interventions — Lacosamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with status epilepticus meets the 2015 diagnostic criteria of the ILAE: Patients with status epilepticus meets the 2015 diagnostic criteria of the International League Against Epilepsy, which is a state in which seizures are persistent and likely to cause long-term impairment, and manifests as:
  1. Tonic-clonic seizures or convulsive seizures, lasting > 5min;
  2. Between 2 or more seizures, consciousness is not restored;
  3. Focal seizures with impaired consciousness, lasting >10min;
  4. absence seizures, lasting > 15min;
  Interventions: Drug: Lacosamide (LCM)

INTERVENTIONS:
Drug: Lacosamide (LCM) — Intravenous lacosamide is given for the treatment of seizure termination in patients with status epilepticus

SUMMARY:
Status epilepticus (SE) is an acute and critical form of neurological and systemic diseases involving multiple clinical disciplines, with an annual incidence of (20-73) per 100,000 people and a clinical case fatality rate of 20%. Although there are many causes of SE, the primary goal of treatment is to terminate the seizures quickly, and timely and standardized treatment can reduce mortality and improve prognosis. The prognosis is closely related to the duration of the episode, and the longer the episode, the worse the prognosis. If seizures of convulsive status epilepticus persist for more than 10 minutes and are not provided with optimal therapeutic intervention, serious adverse outcomes and even death are likely to occur. How to effectively terminate status epilepticus and actively find effective, reliable and safe treatment options is a key research problem at present. Due to critical illness, limited treatment options, and poor prognosis, new treatments are urgently needed to terminate persistent epileptic activity.

Lacosamide (LCM) is a third-generation new antiepileptic drug, which was approved in 2008 for the additive treatment of patients aged 16 years and older with focal seizures, with or without generalized seizures. In 2017, it was extended to patients over 4 years of age. Lacosamide is an anticonvulsant drug with a new dual mechanism of action: first, lacosamide antagonizes the glycine site of N-methyl-D-aspartate (NMDA) receptor; Second, lacosamide selectively acts on the slow inactivation of sodium channels and prolongs the inactivation time of sodium channels, which can more effectively reduce sodium influx and reduce the excitability of neurons, so as to achieve the purpose of treating epilepsy. Lacosamide exhibits linear pharmacokinetics, high oral bioavailability, protein binding of < 15%, rapid and almost complete absorption in a single oral dose, and maximum plasma concentrations within 1 to 4 hours. A number of randomized controlled clinical studies and real-world studies abroad have shown that lacosamide can significantly improve the effective rate and seizure-free rate of epilepsy control, and it is well tolerated and has fewer adverse reactions. The 2022 Chinese Expert Consensus on the Diagnosis and Treatment of Post-stroke Epilepsy recommended lacosamide injection as a first-line drug for non-convulsive status epilepticus after stroke, and the Chinese Expert Consensus on the Diagnosis and Treatment of Status Epilepticus in Children (2022) recommended that lacosamide be considered as an additive treatment for refractory convulsive status epilepticus in children > 60 minutes . There is a lack of clinical research data on the efficacy and safety of intravenous bolus lacosamide for status epilepticus, including convulsive status epilepticus and non-convulsive epilepticus.

DETAILED DESCRIPTION:
In this study, 100 patients with status epilepticus are to be treated. Patients and/or family members signed an informed consent form, and after screening, the participants are enrolled in the group and treated with intravenous lacosamide. The investigators are going to to evaluate the efficacy and safety of intravenous lacosamide in status epilepticus, and to observe the tolerability and adverse effects of lacosamide by observing the seizures and electroencephalogram changes of lacosamide after treatment with lacosamide. All treatments are performed in strict accordance with Good Clinical Practice for Drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 4-60 years old, gender is not limited;
2. Status epilepticus meets the 2015 diagnostic criteria of the International League Against Epilepsy, i.e., a state of persistent seizures that may cause long-term impairment and manifests itself as:

(1) Tonic-clonic seizures or convulsive seizures, lasting > 5min; (2) Between 2 or more seizures, consciousness is not restored; (3) Focal seizures with impaired consciousness, lasting >10min; (4) absence seizures, lasting >15min; 3. Informed consent of the patient and signed a written consent form.

Exclusion Criteria:

1. Unstable vital signs;
2. Electrocardiogram showing atrial flutter, atrial fibrillation, second-degree, third-degree atrioventricular block;
3. History of allergy to the drugs used this time;
4. Participants have a known history of past or present illness of non-epileptic seizures, and current seizures cannot be judged as status epilepticus based on symptomatology and/or electroencephalogram;
5. Other patients who are considered by the investigator to be unsuitable to participate in the study;
6. Incomplete clinical data or follow-up information

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with status epilepticus who are admitted to our hospital and other 4 collaboration hospitals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-06 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Seizure reduction rate | From enrollment to the end of treatment at 1 week
  1. 1-hour status epilepticus termination rate after treatment;
  2. seizure-free rate 24 hours after treatment;
  3. 3 day seizure-free rate after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Na He, Ph.D, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical Universty, Guangzhou, GuanDong, China

IPD SHARING:
Plan to Share IPD: Yes
the efficacy of intravenous lacosamide in the treatment of seizure termination and electroencephalogram improvement in patients with status epilepticus

REFERENCES:
- [Background] Hsiao MR, Tsai TC, Hsia SH, Chan OW, Lee EP, Lin JJ, Lin KL. Intravenous lacosamide for acute repetitive seizures and convulsive status epilepticus in critically ill children. Epilepsia Open. 2024 Dec;9(6):2241-2250. doi: 10.1002/epi4.13047. Epub 2024 Sep 10. PMID 39254674
- [Background] Strzelczyk A, Zollner JP, Willems LM, Jost J, Paule E, Schubert-Bast S, Rosenow F, Bauer S. Lacosamide in status epilepticus: Systematic review of current evidence. Epilepsia. 2017 Jun;58(6):933-950. doi: 10.1111/epi.13716. Epub 2017 Mar 11. PMID 28295226
- [Background] Rogawski MA, Tofighy A, White HS, Matagne A, Wolff C. Current understanding of the mechanism of action of the antiepileptic drug lacosamide. Epilepsy Res. 2015 Feb;110:189-205. doi: 10.1016/j.eplepsyres.2014.11.021. Epub 2014 Dec 3. PMID 25616473
- [Background] Doty P, Rudd GD, Stoehr T, Thomas D. Lacosamide. Neurotherapeutics. 2007 Jan;4(1):145-8. doi: 10.1016/j.nurt.2006.10.002. PMID 17199030
- [Background] Gainza-Lein M, Sanchez Fernandez I, Jackson M, Abend NS, Arya R, Brenton JN, Carpenter JL, Chapman KE, Gaillard WD, Glauser TA, Goldstein JL, Goodkin HP, Kapur K, Mikati MA, Peariso K, Tasker RC, Tchapyjnikov D, Topjian AA, Wainwright MS, Wilfong A, Williams K, Loddenkemper T; Pediatric Status Epilepticus Research Group. Association of Time to Treatment With Short-term Outcomes for Pediatric Patients With Refractory Convulsive Status Epilepticus. JAMA Neurol. 2018 Apr 1;75(4):410-418. doi: 10.1001/jamaneurol.2017.4382. PMID 29356811
- [Background] Coppler PJ, Elmer J. Status Epilepticus: A Neurologic Emergency. Crit Care Clin. 2023 Jan;39(1):87-102. doi: 10.1016/j.ccc.2022.07.006. Epub 2022 Oct 7. PMID 36333039
- [Background] Chin RF, Neville BG, Peckham C, Bedford H, Wade A, Scott RC; NLSTEPSS Collaborative Group. Incidence, cause, and short-term outcome of convulsive status epilepticus in childhood: prospective population-based study. Lancet. 2006 Jul 15;368(9531):222-9. doi: 10.1016/S0140-6736(06)69043-0. PMID 16844492
- [Background] Rossetti AO, Alvarez V. Update on the management of status epilepticus. Curr Opin Neurol. 2021 Apr 1;34(2):172-181. doi: 10.1097/WCO.0000000000000899. PMID 33664203